CLINICAL TRIAL: NCT02178241
Title: Phase II Trial of Gemcitabine-Eribulin (GE) in Cisplatin Ineligible Patients With Advanced or Unresectable Urothelial Carcinoma of the Bladder
Brief Title: Gemcitabine Hydrochloride and Eribulin Mesylate in Treating Patients With Bladder Cancer That is Advanced or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01294; NCI-2014-01294 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P9653_A02PAMDREVW01; PHII-130; 9653 (Other: City of Hope Comprehensive Cancer Center LAO); 9653 (Other: CTEP); N01CM00038 (NIH); P30CA093373 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Ureter Carcinoma; Metastatic Urethral Carcinoma; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7; Stage III Ureter Cancer AJCC v7; Stage III Urethral Cancer AJCC v7; Stage IV Bladder Urothelial Carcinoma AJCC v7; Stage IV Ureter Cancer AJCC v7; Stage IV Urethral Cancer AJCC v7; Ureter Urothelial Carcinoma; Urethral Urothelial Carcinoma
MeSH Terms: conditions — Ureteral Neoplasms; Urethral Neoplasms | interventions — eribulin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (eribulin mesylate and gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011

SUMMARY:
This phase II trial studies how well gemcitabine hydrochloride and eribulin mesylate work in treating patients with bladder cancer that has spread to other places in the body or cannot be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate of gemcitabine (gemcitabine hydrochloride)-eribulin (eribulin mesylate) (GE) when given to cisplatin ineligible patients with advanced or unresectable urothelial carcinoma who have not received any prior chemotherapy for the advanced disease.

SECONDARY OBJECTIVES:

I. To estimate the median progression-free survival (PFS). II. To summarize the toxicity profile (using Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4 criteria) of the GE regimen in these patients.

OUTLINE:

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8 and eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced or metastatic predominantly urothelial carcinoma of the bladder, ureter, or urethra that is not amenable to curative surgical treatment
* Patients must have histologically confirmed predominantly urothelial carcinoma of the bladder, ureter, or urethra
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must be ineligible for treatment with cisplatin, based on one of:

  * Calculated creatinine clearance (CrCl) >= 30 and < 60 mL/min (Cockcroft-Gault)
  * CTCAE grade (Gr) >= 2 hearing loss
  * CTCAE Gr >= 2 neuropathy
* Patients must not have received prior systemic therapy for their advanced cancer; prior intravesical therapy completed 4 weeks prior to enrollment and adjuvant/neoadjuvant chemotherapy completed more than 6 months prior to diagnosis of advanced disease are permitted
* Zubrod performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin < 1.5 times the upper limit of normal (x ULN) for the institution
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine clearance; calculated creatinine clearance (CrCl) >= 30 mL/min and < 60 mL/min (Cockroft-Gault) unless the patient qualified based on hearing loss or neuropathy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of gemcitabine and eribulin administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a small cell component in their histology are excluded
* Patients who have had chemotherapy for the treatment of the advanced or unresectable urothelial cancer of the bladder are not eligible; patients who were previously treated for local disease must not have received radiotherapy or chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study and must have recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have received neoadjuvant or adjuvant chemotherapy must have completed treatment at least 6 months prior to diagnosis of metastatic disease
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine and eribulin
* Uncontrolled intercurrent illness including, but not limited to, a second cancer diagnosis within the past 5 years, or a cancer undergoing any treatment, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with eribulin and gemcitabine
* Human immunodeficiency virus (HIV)-positive patients with inadequate cluster of differentiation (CD)4 counts or those who are on combination antiretroviral therapy with strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) effects are ineligible for this trial
* Patients with baseline corrected QT (QTc) prolongation greater than grade 1 are excluded from this study; patients with grade 1 QTc elevation are eligible but must be monitored with electrocardiogram (ECG) (EKG) exams, for the first 3 cycles of treatment; eribulin time to maximum concentration (Cmax) after infusion is about 10 minutes, and half life is 40 minutes; ECG (EKG) should be performed between 10 to 40 minutes after eribulin administration (on day 1 and day 8 of treatment); continued ECG (EKG) monitoring beyond cycle 3 can be done at the discretion of the treating physician
* Patients with congenital long QT syndrome are excluded from this study
* Other medications known to prolong QT interval should be discontinued and if not possible, patient is excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarmad Sadeghi, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (18):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center P2C, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Mayo Clinic Cancer Center P2C, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas M D Anderson Cancer Center P2C, Houston, Texas
- University Health Network Princess Margaret Cancer Center P2C, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sadeghi S, Groshen SG, Tsao-Wei DD, Parikh R, Mortazavi A, Dorff TB, Kefauver C, Hoimes C, Doyle L, Quinn DI, Newman E, Lara PN Jr. Phase II California Cancer Consortium Trial of Gemcitabine-Eribulin Combination in Cisplatin-Ineligible Patients With Metastatic Urothelial Carcinoma: Final Report (NCI-9653). J Clin Oncol. 2019 Oct 10;37(29):2682-2688. doi: 10.1200/JCO.19.00861. Epub 2019 Aug 7. PMID 31390274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-six patients were enrolled, but 2 did not receive treatment due to medication compliance related to diabetes and another deemed ineligible after registration but prior to treatment start.
Groups:
- Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride): Patients receive 1000mg/m^2 gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and 1.4mg/m^2 eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Eribulin Mesylate: Given IV
  Gemcitabine Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Started (Two enrolled patients did not receive any study treatment and were excluded from analysis.) | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 73 [62 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22
  Hispanic | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Observed Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Observed Overall Response Rate = Number of patients who experienced a confirmed CR or PR divided by the number of eligible patients who began treatment.
Time Frame: Up to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
percentage of participants | 50 [31 to 69]

2. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the start until progression, death, or the start of another treatment, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
months | 5.3 [4.5 to 6.7]

3. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: From start of treatment until death from any cause ,up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
months | 11.9 [5.6 to 20.4]

4. Secondary Outcome: Incidence of Adverse Events.
Description: Toxicities that Occurred in 10% or More of Patients or At Least Once as a Grade 3+ Adverse Event (excluding those toxicities classified as "unrelated" or "unlikely related" to study drugs). Toxicities graded using CTCAEv4 criteria.
Time Frame: Up to 36 months
Measure: Number; unit: participants
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
participants
  Grade 1 or 2 : Anemia | 7
  Grade 1 or 2 : Febrile neutropenia | 3
  Grade 1 or 2 : Thrombotic microangiopathy | 1
  Grade 1 or 2 : Chest pain - cardiac | 0
  Grade 1 or 2 : Heart failure | 0
  Grade 1 or 2 : Colitis | 0
  Grade 1 or 2 : Constipation | 10
  Grade 1 or 2 : Diarrhea | 7
  Grade 1 or 2 : Dry Mouth | 4
  Grade 1 or 2 : Mucositis oral | 2
  Grade 1 or 2 : Nausea | 7
  Grade 1 or 2 : Vomiting | 2
  Grade 1 or 2 : Edema | 9
  Grade 1 or 2 : Fatigue | 13
  Grade 1 or 2 : Fever | 4
  Grade 1 or 2 : Appendicitis perforated | 0
  Grade 1 or 2 : Lung infection | 0
  Grade 1 or 2 : Sepsis | 0
  Grade 1 or 2 : Upper respiratory infection | 0
  Grade 1 or 2 : Urinary Tract Infection | 1
  Grade 1 or 2 : Electrocardiogram QT | 2
  Grade 1 or 2 : Weight Loss | 4
  Grade 1 or 2 : Lymphocyte Count Decreased | 4
  Grade 1 or 2 : Neutrophil Count Decreased | 4
  Grade 1 or 2 : Platelet Count Decreased | 7
  Grade 1 or 2 : White Blood Cell Decreased | 7
  Grade 1 or 2 : INR increased | 1
  Grade 1 or 2 : Alanine Aminotransferase Increased | 9
  Grade 1 or 2 : Aspartate Aminotransferase Incr | 11
  Grade 1 or 2 : Creatinine Increased | 4
  Grade 1 or 2 : Anorexia | 9
  Grade 1 or 2 : Hyperglycemia | 0
  Grade 1 or 2 : Dehydration | 3
  Grade 1 or 2 : Hypoalbuminemia | 8
  Grade 1 or 2 : Hypocalcemia | 4
  Grade 1 or 2 : Hypokalemia | 4
  Grade 1 or 2 : Hypomagnesemia | 3
  Grade 1 or 2 : Hyponatremia | 7
  Grade 1 or 2 : Hypophosphatemia | 4
  Grade 1 or 2 : Generalized Muscle Weakness | 5
  Grade 1 or 2 : Grip Weakness | 0
  Grade 1 or 2 : Pain in Extremity | 3
  Grade 1 or 2 : Dizziness | 5
  Grade 1 or 2 : Dysgeusia | 4
  Grade 1 or 2 : Paresthesia | 4
  Grade 1 or 2 : Peripheral Sensory Neuropathy | 5
  Grade 1 or 2 : Insomnia | 3
  Grade 1 or 2 : Dyspnea | 0
  Grade 1 or 2 : Pneumonitis | 0
  Grade 1 or 2 : Sore Throat | 3
  Grade 1 or 2 : Alopecia | 12
  Grade 1 or 2 : Hypotension | 2
  Grade 1 or 2 : Thromboembolic event | 0
  Grade 3 or 4 : Anemia | 8
  Grade 3 or 4 : Febrile neutropenia | 0
  Grade 3 or 4 : Thrombotic microangiopathy | 0
  Grade 3 or 4 : Chest pain - cardiac | 1
  Grade 3 or 4 : Heart failure | 1
  Grade 3 or 4 : Colitis | 1
  Grade 3 or 4 : Constipation | 0
  Grade 3 or 4 : Diarrhea | 2
  Grade 3 or 4 : Dry Mouth | 0
  Grade 3 or 4 : Mucositis oral | 2
  Grade 3 or 4 : Nausea | 3
  Grade 3 or 4 : Vomiting | 2
  Grade 3 or 4 : Edema | 1
  Grade 3 or 4 : Fatigue | 7
  Grade 3 or 4 : Fever | 0
  Grade 3 or 4 : Appendicitis perforated | 1
  Grade 3 or 4 : Lung infection | 1
  Grade 3 or 4 : Sepsis | 1
  Grade 3 or 4 : Upper respiratory infection | 1
  Grade 3 or 4 : Urinary Tract Infection | 2
  Grade 3 or 4 : Electrocardiogram QT | 1
  Grade 3 or 4 : Weight Loss | 0
  Grade 3 or 4 : Lymphocyte Count Decreased | 6
  Grade 3 or 4 : Neutrophil Count Decreased | 15
  Grade 3 or 4 : Platelet Count Decreased | 3
  Grade 3 or 4 : White Blood Cell Decreased | 13
  Grade 3 or 4 : INR increased | 1
  Grade 3 or 4 : Alanine Aminotransferase Increased | 0
  Grade 3 or 4 : Aspartate Aminotransferase Incr | 1
  Grade 3 or 4 : Creatinine Increased | 0
  Grade 3 or 4 : Anorexia | 0
  Grade 3 or 4 : Hyperglycemia | 1
  Grade 3 or 4 : Dehydration | 2
  Grade 3 or 4 : Hypoalbuminemia | 1
  Grade 3 or 4 : Hypocalcemia | 0
  Grade 3 or 4 : Hypokalemia | 0
  Grade 3 or 4 : Hypomagnesemia | 0
  Grade 3 or 4 : Hyponatremia | 2
  Grade 3 or 4 : Hypophosphatemia | 0
  Grade 3 or 4 : Generalized Muscle Weakness | 1
  Grade 3 or 4 : Grip Weakness | 1
  Grade 3 or 4 : Pain in Extremity | 1
  Grade 3 or 4 : Dizziness | 0
  Grade 3 or 4 : Dysgeusia | 0
  Grade 3 or 4 : Paresthesia | 1
  Grade 3 or 4 : Peripheral Sensory Neuropathy | 0
  Grade 3 or 4 : Insomnia | 0
  Grade 3 or 4 : Dyspnea | 1
  Grade 3 or 4 : Pneumonitis | 1
  Grade 3 or 4 : Sore Throat | 0
  Grade 3 or 4 : Alopecia | 0
  Grade 3 or 4 : Hypotension | 1
  Grade 3 or 4 : Thromboembolic event | 1

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years and 10 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 20/24
Serious Adverse Events (participants affected / at risk) | 16/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride) (N=24)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate and Gemcitabine Hydrochloride) (N=24)
Anemia (Blood and lymphatic system disorders) | 18 (113)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (5)
Blurred vision (Eye disorders) | 2 (5)
Cataract (Eye disorders) | 1 (6)
Dry eye (Eye disorders) | 2 (6)
Watering eyes (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (42)
DUODENITIS (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (16)
Dry mouth (Gastrointestinal disorders) | 4 (16)
Dysphagia (Gastrointestinal disorders) | 3 (5)
Flatulence (Gastrointestinal disorders) | 1 (12)
Gum Bleeding (Gastrointestinal disorders) | 1 (2)
Heartburn (Gastrointestinal disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (13)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 11 (19)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
hematochiza (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 11 (46)
Fatigue (General disorders) | 20 (117)
Fever (General disorders) | 8 (16)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 2 (2)
Injection site reaction (General disorders) | 2 (2)
Leg Pain (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 7 (25)
Plantar fasciitis (General disorders) | 1 (1)
injection site reaction (General disorders) | 1 (1)
vein irritation (General disorders) | 1 (1)
Athlete's foot (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 3 (6)
Toe infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 10 (18)
oral thrush (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (12)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 1 (8)
Alanine aminotransferase increased (Investigations) | 13 (33)
Alkaline phosphatase increased (Investigations) | 6 (16)
Aspartate aminotransferase increased (Investigations) | 12 (42)
Blood bilirubin increased (Investigations) | 2 (5)
Cardiac troponin I increased (Investigations) | 1 (5)
Creatinine increased (Investigations) | 10 (34)
Decreased ANC (Investigations) | 1 (2)
Decreased Creatinine Clearance (Investigations) | 1 (1)
Electrocardiogram QT corrected interval (Investigations) | 3 (8)
INR increased (Investigations) | 4 (21)
Lactic Acidosis Increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 10 (67)
Neutrophil count decreased (Investigations) | 18 (72)
Platelet count decreased (Investigations) | 10 (49)
Weight loss (Investigations) | 4 (14)
White blood cell decreased (Investigations) | 18 (107)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 10 (30)
Decreased eGFR (Metabolism and nutrition disorders) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (65)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (31)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 8 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (15)
Hyponatremia (Metabolism and nutrition disorders) | 10 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (27)
elevated LDH (Metabolism and nutrition disorders) | 1 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (22)
Grip Weakness (Musculoskeletal and connective tissue disorders) | 1 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (12)
grip weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Amnesia (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 5 (25)
Dysgeusia (Nervous system disorders) | 4 (10)
Lethargy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 6 (41)
Peripheral motor neuropathy (Nervous system disorders) | 3 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (28)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (8)
Insomnia (Psychiatric disorders) | 5 (10)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 7 (13)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (3)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (15)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (76)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Erythema RT Lower Leg (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema- RT Lower Leg (Skin and subcutaneous tissue disorders) | 1 (1)
IV site discomfort (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (6)
Purple Macular Lesion Back of Neck (Skin and subcutaneous tissue disorders) | 1 (1)
Purple Macular Lesion Base of Neck (Skin and subcutaneous tissue disorders) | 1 (4)
Purple Macular Leson Base of Neck (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
increased nail growth (Skin and subcutaneous tissue disorders) | 1 (2)
Mediport Placement (Surgical and medical procedures) | 1 (1)
Right Cataract Surgery (Surgical and medical procedures) | 1 (2)
Hypertension (Vascular disorders) | 7 (27)
Hypotension (Vascular disorders) | 3 (9)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02178241/Prot_SAP_000.pdf